CLINICAL TRIAL: NCT03295630
Title: Criterion Validity of the Actigraph GT3X Accelerometer in Determination of Body Position and Walking in Hospital Ward Patients Recovering From Critical Illness
Brief Title: Validity of an Actigraph Accelerometer Following Critical Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R1978
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Critical Care; Walking; Posture
Keywords: Accelerometry; Validity

STUDY DESIGN:
Intervention Model Description: Ankle mounted Actigraph GT3X accelerometer
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Actigraph GT3X accelerometer (Other): Ward based patients recovering from critical illness will wear two accelerometers placed on the thigh and ankle of the non-dominant leg
  Interventions: Device: Accelerometer

INTERVENTIONS:
Device: Accelerometer — Participants will perform a semi-structured movement protocol to investigate the ability of the Actigraph GT3X accelerometer to identify body position (lying, sitting or standing) and quantify step count.

SUMMARY:
This study will determine whether an Actigraph GT3X accelerometer can identify body position and quantify step count in a ward based population recovering from critical illness.

DETAILED DESCRIPTION:
Ward based patients recovering from critical illness who satisfy the inclusion criteria will have an Actigraph GT3X accelerometer positioned on the thigh and ankle of the non dominant leg. These will be used as an objective method of identifying adoption of lying, sitting and standing postures and quantification of step count. Both placement sites will be investigated in isolation. A further analysis will be undertaken to determine whether combining data from both placement sites (ankle and thigh) is superior in identification of lying, sitting and standing postures compared to an isolated single site. Accelerometer data will be compared against direct observation as the criterion measure.

Patients will undertake a semi-structured movement protocol consisting of typical activities undertaken by this population. These include lying in bed, transferring over the side of the bed, sit to stand postural transfers (and the reverse), sitting in a chair and walking. Observation periods will not exceed 3 hours. During this time all aspects of the movement protocol will be completed.

The data from this study will be analysed to determine the validity of the Actigraph GT3X in identification of body position and quantification of step count using the placement sites described above.

ELIGIBILITY:
Inclusion Criteria:

1 18 years of age or above.

2. Ventilated in excess of 48 hours during admission in the Intensive Care Unit (ICU).

3. Currently resident on a hospital ward (secondary care) following step down from ICU

4. Able to undertake all postural transfers independently or with minimal assistance (one person only).

5. Able to mobilise short distances, either independently or with assistance from a walking aid or one person.

6. Willing to permit application of two Actigraph GT3X accelerometers Each device weighs 27g with dimensions of 3.8cm x 3.7cm x 1.8cm.

7. Willing to consent to a period of direct observation for a length of time not exceeding three hours.

Exclusion Criteria:

1. Unable to provide informed written consent themselves
2. Unwilling to consent to a period of observation not exceeding three hours.
3. Unable to make an informed decision about participation or demonstrating an inability to interpret information or follow study instructions
4. Significant neurological or coordination impairment
5. Unable to speak or understand English.
6. Clostridium Difficile/ similar infection or unmanaged urinary incontinence.
7. Evidence/ diagnosis of peripheral vascular disease.
8. Lower limb amputation
9. Polytrauma which prevents the adoption or normal lying, sitting or standing postures, or placement of the accelerometers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2017-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayne Anderson, GradDipPhys, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Hull and East Yorkshire Hospitals NHS Trust, Hull, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 hospital ward based participants recruited. Recruitment period September 2016 to April 2017
Groups:
- Accelerometer (Single Group Recruited): Ward based patients recovering from critical illness will wear two accelerometers placed on the thigh and ankle of the non-dominant leg
  Accelerometer: Participants will perform a semi-structured movement protocol to investigate the ability of the Actigraph GT3X accelerometer to identify body position (lying, sitting or standing) and quantify step count
Period: Overall Study
Arm/Group | Accelerometer (Single Group Recruited)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Accelerometer: Ward based patients recovering from critical illness will wear two accelerometers placed on the thigh and ankle of the non-dominant leg
  Accelerometer: Participants will perform a semi-structured movement protocol to investigate the ability of the Actigraph GT3X accelerometer to identify body position (lying, sitting or standing) and quantify step count
Arm/Group | Accelerometer
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Years]
  United Kingdom | 20
Gender [Count of Participants; unit: Participants]
  Male | 13
  Female | 7
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.9 (6.1)
Number of days receiving mechanical ventilation [Median (Inter-Quartile Range); unit: days] | 15 [5.5 to 36]
ICU overall length of stay [Median (Inter-Quartile Range); unit: days] | 21 [8.25 to 42.75]
Overall hospital length of stay [Median (Inter-Quartile Range); unit: days] | 35 [17.25 to 64.75]

OUTCOME MEASURES:

1. Primary Outcome: Ability of an Accelerometer to Identify Step Count
Description: Agreement between direct observation and the activity monitors (ankle and thigh placements in isolation) in determination of step count. The mean difference (95% Limits of Agreement) between observed step count and accelerometer quantified step count for the same walk were calculated. Negative values reflected an underestimation of observed step count by the accelerometer and positive values reflected an overestimation of step count.
Time Frame: Participants wore the accelerometers for a maximum of 3 hours, undertaking a semi-structured movement protocol
Population: Investigation of agreement between accelerometer quantified step count (ankle and thigh in isolation) and observed step count
Measure: Mean (Full Range); unit: Observed steps
Arm/Group | Accelerometer
Number analyzed (Participants) | 20
Observed steps | 46 [15 to 90]
Statistical Analysis 1: Comparison: Accelerometer; Difference (steps) between accelerometer quantified step count (thigh placement) and observed step count; Test type: Other; Mean Difference (Final Values) = -17.7
Statistical Analysis 2: Comparison: Accelerometer; Correlation between accelerometer quantified step count (thigh placement) and observed step count; Test type: Other; Intraclass Correlation Coefficient = 0.46, 95% CI 2-sided [-0.1 to 0.78]
Statistical Analysis 3: Comparison: Accelerometer; Difference (steps) between accelerometer quantified steps (ankle placement) and observed step count; Test type: Other; Mean Difference (Final Values) = -0.84
Statistical Analysis 4: Comparison: Accelerometer; Correlation between accelerometer quantified steps (ankle placement) and observed steps; Test type: Other; Intraclass Correlation Coefficient = 0.99, 95% CI 2-sided [0.99 to 1.0]

2. Secondary Outcome: Comfort of Accelerometers
Description: Participants were asked to rate their assessment of how comfortable the accelerometers were. They were requested to choose a statement on a five-point Likert Scale. The statements were:
  1. Very uncomfortable
  2. Somewhat uncomfortable
  3. Neither comfortable nor uncomfortable
  4. Somewhat comfortable
  5. Very comfortable
  Participants chose the most appropriate statement which they felt reflected how comfortable they found the accelerometers to wear.
Time Frame: Accelerometers were worn for a period not exceeding 3 hours
Population: Participants were asked to rate accelerometer comfort using a 5-point Likert Scale with the following statements:
  'Very comfortable', 'Somewhat comfortable', 'Neither comfortable or uncomfortable', Somewhat uncomfortable', Very uncomfortable'
Measure: Count of Participants; unit: Participants
Groups:
- Accelerometer: Participants rating of accelerometer comfort using a 5-point Likert Scale
Arm/Group | Accelerometer
Number analyzed (Participants) | 20
Participants
  Very Comfortable | 16
  Somewhat comfortable | 3
  Neither comfortable or uncomfortable | 0
  Somewhat uncomfortable | 1
  Very uncomfortable | 0

ADVERSE EVENTS:
Time Frame: Not exceeding 3 hours
Arm/Group | Accelerometer (Single Group Recruited)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT03295630/Prot_SAP_000.pdf
  • Informed Consent Form (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT03295630/ICF_001.pdf